CLINICAL TRIAL: NCT05846867
Title: An Open, Multicenter Phase Ib/II Clinical Study on the Efficacy and Safety of AK119 and AK112, Either in Combination or Not, With Chemotherapy, and AK112 Monotherapy in pMMR/MSS CRC
Brief Title: A Phase Ib/II Clinical Study on AK112 Combined or Not Combined With AK119 in pMMR/MSS Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK119-202
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- AK119 20mg/kg+ AK112 20mg/kg (Experimental): Subjects will receive AK119 plus AK112 via intravenously (IV) Q2W, up to 2 years
  Interventions: Drug: AK119; Drug: AK112
- AK119 40mg/kg+ AK112 20mg/kg (Experimental): Subjects will receive AK119 plus AK112 via intravenously (IV) Q2W, up to 2 years
  Interventions: Drug: AK119; Drug: AK112
- AK119 + AK112 20mg/kg +mFOLFOX6 (Experimental): Subjects will receive AK119 and AK112 plus mFOLFOX6 via intravenously (IV)Q2W, up to 12 cycles. Afterward, AK119 and AK112 will continue to be treated up to 2 years.
  Interventions: Drug: AK119; Drug: AK112; Drug: Oxaliplatin; Drug: Calcium folinate; Drug: Fluorouracil
- AK119 + AK112 20mg/kg +FOLFIRI (Experimental): Subjects will receive AK119 and AK112 plus FOLFIRI via intravenously (IV)Q2W, up to 12 cycles. Afterward, AK119 and AK112 will continue to be treated up to 2 years.
  Interventions: Drug: AK119; Drug: AK112; Drug: Irinotecan; Drug: Calcium folinate; Drug: Fluorouracil
- AK112 20mg/kg (Experimental): Subjects will receive AK112 via intravenously (IV) Q2W, up to 2 years
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK119 — AK119 IV every 2 weeks.intravenous infusion
  Arms: AK119 + AK112 20mg/kg +FOLFIRI; AK119 + AK112 20mg/kg +mFOLFOX6; AK119 20mg/kg+ AK112 20mg/kg; AK119 40mg/kg+ AK112 20mg/kg
Drug: AK112 — AK112 IV every 2 weeks.intravenous infusion
Drug: Oxaliplatin — Oxaliplatin: 85mg/m2, intravenous infusion
  Arms: AK119 + AK112 20mg/kg +mFOLFOX6
Drug: Irinotecan — Irinotecan 180mg/m2, intravenous infusion
  Arms: AK119 + AK112 20mg/kg +FOLFIRI
Drug: Calcium folinate — Calcium folinate: 400mg/m2, intravenous infusion
  Arms: AK119 + AK112 20mg/kg +FOLFIRI; AK119 + AK112 20mg/kg +mFOLFOX6
Drug: Fluorouracil — Fluorouracil 400mg/m2, intravenous injection
  Arms: AK119 + AK112 20mg/kg +FOLFIRI; AK119 + AK112 20mg/kg +mFOLFOX6

SUMMARY:
This is an open label, multicenter Phase Ib/II clinical study on the efficacy and safety of AK119 and AK112 in combination with or without chemotherapy, and AK112 monotherapy in pMMR/MSS CRC

DETAILED DESCRIPTION:
This study is an open, multicenter, Ib/II phase clinical trial conducted in China. The research plan is divided into 5 queues. A total of 130-170 subjects were enrolled. Subjects who meet the research criteria will receive treatment with AK119 and AK112 in combination or without chemotherapy, as well as AK112 monotherapy, every two weeks according to the protocol. The research on the first and second cohorts will be conducted first, and at least two lines of microsatellite stabilized colorectal cancer subjects who have failed standard treatment will be enrolled; Subsequently, a third cohort was conducted, which included microsatellite stabilized colorectal cancer subjects who had failed at least two lines of standard treatment; After preliminary confirmation of the safety and efficacy of AK119 combined with AK112 in the first and second cohorts, and determination of the recommended dose of AK119 for subsequent combination chemotherapy, the study of AK119 and AK112 combined chemotherapy in the fourth and fifth cohorts will be conducted. The fourth and fifth cohorts will include participants with advanced first-line microsatellite stable colorectal cancer who have not received systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and voluntarily sign the written informed consent, which must be signed before the specified research procedure required by the research is implemented.
2. Age ≥ 18 when signing the informed consent form (ICF), both male and female。
3. Microsatellite stable colorectal cancer confirmed by histopathology; Microsatellite stability was defined as the expression of four common MMR proteins (MLH1, MSH2, MSH6 and PMS2) detected by immunohistochemistry, and all four proteins were positive for pMMR. Or PCR method was used to detect sites (BAT25, BAT26, D5S346, D2S123 and D17S250), and the detection results showed that the stability was microsatellite stability or microsatellite low degree instability.
4. The first and second cohorts: recurrent or metastatic colorectal cancer that has failed to undergo at least the second-line standard treatment in the past; The chemotherapy of at least one of the treatment lines is the combination chemotherapy of at least two cytotoxic drugs based on platinum or irinotecan; Definition of treatment failure: disease progression occurs during or after treatment. All patients who change the treatment plan due to drug intolerance are not considered as treatment failure; For subjects who have received induction chemotherapy, concurrent radiotherapy and chemotherapy or adjuvant chemotherapy in the past, if relapse/metastasis occurs within 6 months after the last treatment, the original treatment plan is defined as the first-line treatment plan for the subject.
5. The third and fourth cohorts: for patients with advanced colorectal cancer who have not undergone systematic treatment, the recurrence time should be at least 6 months from the end of the last treatment for those who have previously received induction chemotherapy, concurrent radiotherapy and chemotherapy or adjuvant/neoadjuvant chemotherapy.
6. Agree to provide archived or freshly obtained tumor tissue samples within 2 years before the first administration (preferably newly obtained tumor tissue samples) About 20 unstained FFPE pathological sections (if the sample size is not enough, only 10 unstained FFPE pathological sections can be provided with the approval of medical inspectors FFPE pathological section).
7. According to RECIST v1.1 standard, subjects have at least one measurable target lesion; The focus that has received radiotherapy is not selected as the target lesion, unless the radiotherapy focus is the only measurable focus and the progress is determined according to the imaging, it can be considered as the target lesion.
8. The Eastern Cancer Cooperation Organization (ECOG) physical state score is 0 or 1.
9. The expected survival period is ≥ 3 months.

Exclusion Criteria:

1. Pathological examination confirmed other pathological types, such as squamous cell carcinoma, sarcoma or undifferentiated carcinoma, gastrointestinal stromal tumor, etc.
2. Palliative local treatment for non-target lesions within 2 weeks before the first administration; Have received systemic non-specific immunomodulation therapy (such as interleukin, interferon, thymosin, etc.) within 2 weeks before the first administration; Received Chinese herbal medicine or traditional Chinese patent medicines and simple preparations with anti-tumor indications within 2 weeks before the first administration。
3. Had been treated with anti-CD73 inhibitors, immune checkpoint inhibitors (such as anti-PD-1 antibody, anti-PD-L1 antibody, anti-CTLA-4 antibody, etc.), immune checkpoint agonists (such as antibodies against ICOS, CD40, CD137, GITR, OX40 targets, etc.), immune cell therapy (such as CAR-T) and other therapies aimed at tumor immune mechanism.
4. There is a history of gastrointestinal perforation and fistula within 6 months before the first administration. If the perforation or fistula has been removed or repaired, and the researcher judges that the disease has recovered or alleviated, it can be admitted into the group.
5. Active or inactive Inflammatory bowel disease (such as Crohn's disease or ulcerative colitis) previously recorded. Inability to swallow, malabsorption syndrome, or uncontrollable nausea, vomiting, diarrhea or other gastrointestinal diseases that seriously affect the use and absorption of drugs.
6. Except for the tumor that the subject had at the time of enrollment, there was active malignant tumor in the previous five years. However, the tumors participating in the study and cured local tumors are excluded, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, breast carcinoma in situ, localized prostate cancer, etc.
7. At the same time, another interventional clinical study was enrolled.
8. Receive the last systemic anti-tumor treatment within 3 weeks before the first administration; Received small molecular TKI treatment within 2 weeks before the first administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or confirmed PR
Number of subjects with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of study drug
  AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.
recommended phaseII dose | 1 year
  Phase II clinical study recommended dose (RP2D) of AK119 and AK112 combined with or without chemotherapy

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST Version 1.1)
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (based on RECIST Version 1.1).
Duration of response (DoR) | Up to 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST Version 1.1) or death due to any cause, whichever occurs first
Time to response (TTR) | Up to 2 years
  TTR is defined as the time from the start of the treatment to the first objective tumor response observed for patients who achieved CR or PR (based on RECIST Version 1.1)
Total survival time (OS) and 12-month OS rate | Up to 2 years
  OS defined as the time from the first dose to death from any cause
Maximum observed concentration (Cmax) of AK119 and AK112 | From first dose of study drug through last dose up to 100 weeks
  The PK parameters include serum concentrations of AK119 and AK112 at different timepoints after study drug administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of study drug through last dose up to 100 weeks
  The immunogenicity of AK119 and AK112 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).
Correlation between biomarkers and efficacy | Up to 2 years
  Correlation between the expression level of PD-L1 and CD73 biomarkers and efficacy ORR, PFS and OS

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiao Zhang, PhD, Study Chair — Cancer Hospital Affiliated to Harbin Medical University
Locations (1):
- Cancer Hospital Affiliated to Harbin Medical University, Harbin, China

IPD SHARING:
Plan to Share IPD: No